CLINICAL TRIAL: NCT04305353
Title: Implementing an Intensive Care Unit (ICU) Diary Program at a Large Academic Medical Center: Results From a Randomized Control Trial Evaluating Psychological Morbidity Associated With Critical Illness
Brief Title: Intensive Care Unit (ICU) Diary Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tulane University School of Medicine (Other)
Collaborators: The Arnold P. Gold Foundation (Other)
Responsible Party: Sponsor
Organization: Tulane University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ICU Diary RCT NOLA; GH-17-022 (Other Grant/Funding Number: The Arnold P. Gold Foundation)
Record Dates: First submitted 2020-02-13; First posted 2020-03-12 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: PTSD; Post ICU Syndrome
Keywords: psychocognitive morbidity; narrative medicine; ICU-related PTSD; Post-ICU Syndrome (PICS); ICU Diary
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Narrative Medicine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ICU Diary Group (Experimental): Patients randomized to this group receive the ICU diary, along with PTSD education
  Interventions: Other: Diary (blank journal) plus PTSD psycho-education; Other: PTSD psycho-education alone
- PTSD Education-only Group (Other): Control Group: patients randomized to this group only receive PTSD education
  Interventions: Other: PTSD psycho-education alone

INTERVENTIONS:
Other: Diary (blank journal) plus PTSD psycho-education — A blank journal where a prospective account of a patient's ICU course (everyday events) can be documented by family members and healthcare providers
  Arms: ICU Diary Group
Other: PTSD psycho-education alone — We administered a pamphlet to patients with information regarding PTSD symptoms, potential psychiatric complications after discharge, and available mental health resources.
  References for our education include the following which are included in our references section: Jensen 2015, Jones 2010, Knowles 2009, Parker 2015, Wintermann 2015.

SUMMARY:
Psychological morbidity in both patients and family members related to the intensive care unit (ICU) experience is an often overlooked, and potentially persistent, healthcare problem recognized by the Society of Critical Care Medicine as Post-intensive Care Syndrome (PICS). ICU diaries are an intervention increasingly under study with potential to mitigate ICU-related psychological morbidity, include ICU-related PTSD (post-traumatic stress disorder), depression and anxiety.

DETAILED DESCRIPTION:
The investigators compared the efficacy of the ICU diary, prospectively written by third-parties during the patient's intensive care course, versus education-alone, on reducing acute PTSD symptoms after discharge. Patients with an ICU stay greater than 72 hours, and who were intubated and mechanically ventilated over 24 hours, were recruited and randomized to either receive a diary at bedside with psychoeducation, or psychoeducation alone. Intervention patients received their ICU diary within the first week of admission into the intensive care unit. Psychometric testing with IES-R, PHQ-8, HADS and GAD-7 was conducted at weeks 4, 12, and 24 after ICU discharge.

ELIGIBILITY:
Inclusion Criteria:

* admitted to the intensive care unit for at least 72 hours
* sedated and mechanically ventilated for at least 24 hours.
* available over-the-phone, up to 6 months post-ICU discharge

Exclusion Criteria:

* any patients who do not voluntarily agree to participate
* not fluent in the English language
* patients who have stayed in the ICU for less than 72 hours
* patients who have been sedated and mechanically ventilated for less than 24 hours
* patients with pre-existing severe psychotic illness, bipolar disorder, substance use disorder, PTSD, stroke, traumatic brain injury, neurocognitive impairment, or intellectual disability
* patients with no phone number or reliable contact information for the sake of follow-up
* prisoners
* pregnant patients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-09-26 (Actual); Primary Completion 2018-09-25 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Change in PTSD symptoms | at baseline (within one week of ICU admission) versus twelve-weeks post-ICU discharge
  Revised Impact of Event Scales (IES-R) score, measuring areas of hyperarousal, avoidance, and intrusion as subscales. Total score ranges from 0-88, higher score associated with worse PTSD symptoms. Scores from 1-22 are consistent with mild PTSD, and scores greater than 22 signal clinically significant PTSD symptoms.

SECONDARY OUTCOMES:
Change in Hospital-associated Depression and Anxiety symptoms | at baseline (within one week of ICU admission) versus twelve-weeks post-ICU discharge
  Hospital Anxiety and Depression Scale (HADS), range of 0-21 for either anxiety or depression subscores, with higher scores corresponding to worse outcomes. Scores of 0-7 are normal, 8-10 are borderline abnormal (mild depression or anxiety), and 11-21 correspond to severe symptoms of anxiety or depression.
Change in Depression symptoms | at baseline (within one week of ICU admission) versus twelve-weeks post-ICU discharge
  Patient Health Questionnaire (PHQ-8), score ranges 0-24, as higher scores correspond to worse depression symptoms. Scores of 5-10 represent mild symptoms of depression, 10-15 signal moderate symptoms, and 15-24 correspond to severe symptoms.
Change in Anxiety symptoms | at baseline (within one week of ICU admission) versus twelve-weeks post-ICU discharge
  Generalized Anxiety Disorder 7-item scores (GAD-7) range from 0 to 21, with higher scores corresponding to worse anxiety symptoms. Scores of 0-4 indicate minimal anxiety, 5-9 correspond to mild anxiety, 10-14 signal moderate anxiety, and 15-21 represent severe anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Hammer, MD, MFA, Principal Investigator — Tulane University School of Medicine; George Sayde, MD, MPH, Principal Investigator — Tulane University School of Medicine
Locations (1):
- Tulane University School of Medicine, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Parker AM, Sricharoenchai T, Raparla S, Schneck KW, Bienvenu OJ, Needham DM. Posttraumatic stress disorder in critical illness survivors: a metaanalysis. Crit Care Med. 2015 May;43(5):1121-9. doi: 10.1097/CCM.0000000000000882. PMID 25654178
- [Background] Wintermann GB, Brunkhorst FM, Petrowski K, Strauss B, Oehmichen F, Pohl M, Rosendahl J. Stress disorders following prolonged critical illness in survivors of severe sepsis. Crit Care Med. 2015 Jun;43(6):1213-22. doi: 10.1097/CCM.0000000000000936. PMID 25760659
- [Background] Jones C, Backman C, Capuzzo M, Egerod I, Flaatten H, Granja C, Rylander C, Griffiths RD; RACHEL group. Intensive care diaries reduce new onset post traumatic stress disorder following critical illness: a randomised, controlled trial. Crit Care. 2010;14(5):R168. doi: 10.1186/cc9260. Epub 2010 Sep 15. PMID 20843344
- [Background] Myhren H, Ekeberg O, Toien K, Karlsson S, Stokland O. Posttraumatic stress, anxiety and depression symptoms in patients during the first year post intensive care unit discharge. Crit Care. 2010;14(1):R14. doi: 10.1186/cc8870. Epub 2010 Feb 8. PMID 20144193
- [Background] Jensen JF, Thomsen T, Overgaard D, Bestle MH, Christensen D, Egerod I. Erratum to: Impact of follow-up consultations for ICU survivors on post-ICU syndrome: a systematic review and meta-analysis. Intensive Care Med. 2015 Jul;41(7):1391. doi: 10.1007/s00134-015-3932-9. No abstract available. PMID 26104120
- [Background] Davydow DS, Kohen R, Hough CL, Tracy JH, Zatzick D, Katon WJ. A pilot investigation of the association of genetic polymorphisms regulating corticotrophin-releasing hormone with posttraumatic stress and depressive symptoms in medical-surgical intensive care unit survivors. J Crit Care. 2014 Feb;29(1):101-6. doi: 10.1016/j.jcrc.2013.08.016. Epub 2013 Sep 24. PMID 24075295
- [Background] Jones C, Backman C, Griffiths RD. Intensive care diaries and relatives' symptoms of posttraumatic stress disorder after critical illness: a pilot study. Am J Crit Care. 2012 May;21(3):172-6. doi: 10.4037/ajcc2012569. PMID 22549573
- [Background] Knowles RE, Tarrier N. Evaluation of the effect of prospective patient diaries on emotional well-being in intensive care unit survivors: a randomized controlled trial. Crit Care Med. 2009 Jan;37(1):184-91. doi: 10.1097/CCM.0b013e31819287f7. PMID 19050634
- [Background] Jones C, Griffiths RD, Humphris G, Skirrow PM. Memory, delusions, and the development of acute posttraumatic stress disorder-related symptoms after intensive care. Crit Care Med. 2001 Mar;29(3):573-80. doi: 10.1097/00003246-200103000-00019. PMID 11373423
- [Background] Karnatovskaia LV, Johnson MM, Benzo RP, Gajic O. The spectrum of psychocognitive morbidity in the critically ill: a review of the literature and call for improvement. J Crit Care. 2015 Feb;30(1):130-7. doi: 10.1016/j.jcrc.2014.09.024. Epub 2014 Oct 2. PMID 25449881
- [Background] Bergbom I, Svensson C, Berggren E, Kamsula M. Patients' and relatives' opinions and feelings about diaries kept by nurses in an intensive care unit: pilot study. Intensive Crit Care Nurs. 1999 Aug;15(4):185-91. doi: 10.1016/s0964-3397(99)80069-x. PMID 10786503
- [Background] Ullman AJ, Aitken LM, Rattray J, Kenardy J, Le Brocque R, MacGillivray S, Hull AM. Diaries for recovery from critical illness. Cochrane Database Syst Rev. 2014 Dec 9;2014(12):CD010468. doi: 10.1002/14651858.CD010468.pub2. PMID 25488158
- [Background] Garrouste-Orgeas M, Flahault C, Vinatier I, Rigaud JP, Thieulot-Rolin N, Mercier E, Rouget A, Grand H, Lesieur O, Tamion F, Hamidfar R, Renault A, Parmentier-Decrucq E, Monseau Y, Argaud L, Bretonniere C, Lautrette A, Badie J, Boulet E, Floccard B, Forceville X, Kipnis E, Soufir L, Valade S, Bige N, Gaffinel A, Hamzaoui O, Simon G, Thirion M, Bouadma L, Large A, Mira JP, Amdjar-Badidi N, Jourdain M, Jost PH, Maxime V, Santoli F, Ruckly S, Vioulac C, Leborgne MA, Bellalou L, Fasse L, Misset B, Bailly S, Timsit JF. Effect of an ICU Diary on Posttraumatic Stress Disorder Symptoms Among Patients Receiving Mechanical Ventilation: A Randomized Clinical Trial. JAMA. 2019 Jul 16;322(3):229-239. doi: 10.1001/jama.2019.9058. PMID 31310299
- [Derived] Sayde GE, Stefanescu A, Conrad E, Nielsen N, Hammer R. Implementing an intensive care unit (ICU) diary program at a large academic medical center: Results from a randomized control trial evaluating psychological morbidity associated with critical illness. Gen Hosp Psychiatry. 2020 Sep-Oct;66:96-102. doi: 10.1016/j.genhosppsych.2020.06.017. Epub 2020 Jul 2. PMID 32763640